CLINICAL TRIAL: NCT01318122
Title: A Long-Term, Open-Label Extension Study to Investigate the Long-Term Safety of SYR-322 When Used in Combination With Thiazolidine in Subjects With Type 2 Diabetes in Japan
Brief Title: Long-term Safety Study of Alogliptin Used in Combination With Thiazolidine in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322/OCT-004; U1111-1119-6207 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD (Active Comparator)
  Interventions: Drug: Alogliptin and pioglitazone
- Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (Active Comparator)
  Interventions: Drug: Alogliptin and pioglitazone

INTERVENTIONS:
Drug: Alogliptin and pioglitazone — Alogliptin 12.5 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322; Actos
  Arms: Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD
Drug: Alogliptin and pioglitazone — Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  Other Names: SYR-322; Actos
  Arms: Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD

SUMMARY:
The purpose of this study was to evaluate the long-term safety and efficacy of alogliptin and Thiazolidine administered once daily (QD) for 40 consecutive weeks in participants who completed a phase 2/3 Thiazolidine add on study.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

To evaluate the long-term safety and efficacy of alogliptin, participants in the present study were enrolled from a core phase 2/3 thiazolidine add on study (SYR-322/CCT-004; NCT01318070).

ELIGIBILITY:
Inclusion Criteria:

1. Had completed the core phase 2/3 thiazolidine add on study.
2. The subject was capable of understanding and complying with protocol requirements.
3. Signed a written, informed consent form prior to the initiation of any study procedure.

Exclusion Criteria:

1. With clinical manifestation of hepatic impairment (e.g., an AST or ALT value of 2.5 times or more of the upper reference limit at Week 8 of the core phase 2/3 thiazolidine add on study).
2. With clinical manifestation of renal impairment (e.g., a creatinine value of 2 mg/dL or more at Week 8 of the core phase 2/3 thiazolidine add on study).
3. With a history or symptoms of cardiac failure.

Ages: 33 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Department of Medicine, Study Director — Department of Medicine, Kawasaki Medical School

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 32 investigative sites in Japan from 10 May 2008 to 03 August 2009.
Pre-assignment Details: Participants who had completed the core phase 2/3 thiazolidine add on study (SYR-322/CCT-004; NCT01318070) were enrolled in one of 2, once-daily (QD) treatment groups.
Groups:
- CCT/004 - 12.5 mg Dose Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  *for participants from the 12.5 mg combination dosing ARM of the SYR-322/CCT-004 (NCT01318070) core phase 2/3 pioglitazone add-on study.
- CCT/004 - 25 mg Dose Group* → 25 mg Combination Dose Group: Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  *for participants from the 25 mg combination dosing ARM of the SYR-322/CCT-004 (NCT01318070) core phase 2/3 pioglitazone add-on study.
- Pioglitazone Monotherapy Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  *for participants from the pioglitazone 15 mg or 30 mg dosing ARM of the SYR-322/CCT-004 (NCT01318070) core phase 2/3 pioglitazone add-on study.
- Pioglitazone Monotherapy Group* → 25 mg Combination Group: Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  *for participants from the pioglitazone 15 mg or 30 mg dosing ARM of the SYR-322/CCT-004 (NCT01318070) core phase 2/3 pioglitazone add-on study.
Period: Enrolled - Long-Term Extension Study
Arm/Group | CCT/004 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/004 - 25 mg Dose Group* → 25 mg Combination Dose Group | Pioglitazone Monotherapy Group* → 12.5 mg Combination Group | Pioglitazone Monotherapy Group* → 25 mg Combination Group
Started | 106 (5 randomized participants from alogliptin 12.5 & 25 mg group CCT-004 study did not enter this study) | 110 (5 randomized participants from alogliptin 12.5 & 25 mg group CCT-004 study did not enter this study) | 57 | 53
Completed | 105 | 110 | 55 | 52
Not Completed | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 1
Not completed — Other | 1 | 0 | 0 | 0
Period: Entered - Long-Term Extension Study
Arm/Group | CCT/004 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/004 - 25 mg Dose Group* → 25 mg Combination Dose Group | Pioglitazone Monotherapy Group* → 12.5 mg Combination Group | Pioglitazone Monotherapy Group* → 25 mg Combination Group
Started | 105 | 110 | 55 | 52
Completed | 96 | 99 | 49 | 48
Not Completed | 9 | 11 | 6 | 4
Not completed — Adverse Event | 6 | 6 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
- Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD: Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD | Total
Number analyzed (Participants) | 166 | 165 | 331
Age, Customized [Number; unit: participants]
  ≤ 64 years | 116 | 103 | 219
  ≥ 65 years | 50 | 62 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 58 | 123
  Male | 101 | 107 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: Treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Time Frame: 52 Weeks.
Population: Full Analysis Set was defined as the population of participants randomized in the core phase 2/3 thiazolidine add on study (SYR-322/CCT-004 study; NCT01318070) and received at least 1 dose of the investigational products (SYR-322DB in combination with pioglitazone) for the treatment period.
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 166 | 165
participants
  Number of Participants with Serious Adverse Event | 14 | 11
  Number of Participants with Other Adverse Event | 143 | 146

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 165 | 164
percentage of Glycosylated Hemoglobin | -0.68 (0.371) | -0.73 (0.415)

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 161 | 163
percentage of Glycosylated Hemoglobin | -0.81 (0.459) | -0.88 (0.519)

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 158 | 160
percentage of Glycosylated Hemoglobin | -0.86 (0.550) | -0.92 (0.571)

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 155 | 160
percentage of Glycosylated Hemoglobin | -0.84 (0.616) | -0.90 (0.581)

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 24).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 155 | 158
percentage of Glycosylated Hemoglobin | -0.78 (0.612) | -0.82 (0.585)

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 28).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 28 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 151 | 156
percentage of Glycosylated Hemoglobin | -0.75 (0.620) | -0.76 (0.597)

8. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 32).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 32 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 150 | 152
percentage of Glycosylated Hemoglobin | -0.72 (0.605) | -0.72 (0.632)

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 36).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 36 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 147 | 151
percentage of Glycosylated Hemoglobin | -0.67 (0.575) | -0.69 (0.599)

10. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 40).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 40 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 147 | 150
percentage of Glycosylated Hemoglobin | -0.65 (0.573) | -0.66 (0.603)

11. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 44).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 44 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 98 | 101
percentage of Glycosylated Hemoglobin | -0.70 (0.577) | -0.74 (0.629)

12. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 48).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 48 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 98 | 101
percentage of Glycosylated Hemoglobin | -0.73 (0.596) | -0.76 (0.683)

13. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 52).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 96 | 100
percentage of Glycosylated Hemoglobin | -0.77 (0.571) | -0.79 (0.633)

14. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Final Visit).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 166 | 165
percentage of Glycosylated Hemoglobin | -0.65 (0.597) | -0.65 (0.659)

15. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 8).
Description: The change between the value of fasting blood glucose collected at week 8 and baseline.
Time Frame: Baseline and Week 8.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 165 | 164
mg/dL | -15.5 (19.60) | -18.1 (20.82)

16. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 12).
Description: The change between the value of fasting blood glucose collected at week 12 and baseline.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 161 | 163
mg/dL | -13.4 (18.37) | -16.3 (20.54)

17. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 16).
Description: The change between the value of fasting blood glucose collected at week 6 and baseline.
Time Frame: Baseline and Week 16.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 158 | 160
mg/dL | -11.9 (22.04) | -13.4 (20.81)

18. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 20).
Description: The change between the value of fasting blood glucose collected at week 20 and baseline.
Time Frame: Baseline and Week 20.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 155 | 160
mg/dL | -10.1 (21.07) | -13.9 (21.74)

19. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 24).
Description: The change between the value of fasting blood glucose collected at week 24 and baseline.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 155 | 158
mg/dL | -10.0 (21.50) | -10.7 (23.02)

20. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 28).
Description: The change between the value of fasting blood glucose collected at week 28 and baseline.
Time Frame: Baseline and Week 28.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 151 | 156
mg/dL | -5.6 (28.42) | -9.1 (21.27)

21. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 32).
Description: The change between the value of fasting blood glucose collected at week 32 and baseline.
Time Frame: Baseline and Week 32.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 150 | 152
mg/dL | -7.9 (20.25) | -10.4 (21.27)

22. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 36).
Description: The change between the value of fasting blood glucose collected at week 36 and baseline.
Time Frame: Baseline and Week 36.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 147 | 151
mg/dL | -7.1 (19.65) | -11.9 (18.33)

23. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 40).
Description: The change between the value of fasting blood glucose collected at week 40 and baseline.
Time Frame: Baseline and Week 40.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 147 | 150
mg/dL | -9.5 (20.76) | -10.6 (27.38)

24. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 44).
Description: The change between the value of fasting blood glucose collected at week 44 and baseline.
Time Frame: Baseline and Week 44.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 98 | 101
mg/dL | -10.4 (17.43) | -10.4 (21.24)

25. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 48).
Description: The change between the value of fasting blood glucose collected at week 48 and baseline.
Time Frame: Baseline and Week 48.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 98 | 101
mg/dL | -12.2 (19.89) | -14.0 (21.91)

26. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 52).
Description: The change between the value of fasting blood glucose collected at week 52 and baseline.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 96 | 100
mg/dL | -12.8 (16.63) | -13.6 (26.28)

27. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Final Visit).
Description: The change between the value of fasting blood glucose collected at week 52 or final visit and baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 166 | 165
mg/dL | -11.4 (19.29) | -11.1 (25.19)

28. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 12).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 12 and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 163 | 163
mg/dL | 58.3 (30.81) | 49.5 (30.04)

29. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 24).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 24 and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 104 | 109
mg/dL | 55.9 (30.87) | 47.9 (29.20)

30. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 52).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 52 or final visit and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 146 | 147
mg/dL | 59.1 (34.19) | 57.2 (31.82)

31. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Final Visit).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 52 or end of study and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Number analyzed (Participants) | 163 | 163
mg/dL | 59.8 (34.26) | 56.8 (32.12)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through receiving the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. 5 participants from alogliptin 12.5 & 25 mg group CCT-004 study did not enter this study.
Groups:
- Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD: Alogliptin 25 mg, tablets, orally, once daily and Pioglitazone 15 mg or 30 mg, tablets, orally, once daily for up to 40 weeks.
  *for participants from the 25 mg combination dosing ARM of the SYR-322/CCT-004 (NCT01318070) core phase 2/3 pioglitazone add-on study.
Arm/Group | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD
Serious Adverse Events (participants affected / at risk) | 14/166 | 11/165
Other Adverse Events (participants affected / at risk) | 143/166 | 146/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD (N=166) | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (N=165)
Epiglottitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cataract (Eye disorders) | 1 | 3
Diabetic retinopathy (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Pioglitazone 15 or 30 mg QD (N=166) | Alogliptin 25 mg QD and Pioglitazone 15 or 30 mg QD (N=165)
Nasopharyngitis (Infections and infestations) | 54 | 54
Bronchitis (Infections and infestations) | 8 | 2
Pharyngitis (Infections and infestations) | 4 | 6
Headache (Nervous system disorders) | 5 | 6
Diabetic retinopathy (Eye disorders) | 7 | 6
Conjunctivitis allergic (Eye disorders) | 1 | 5
Hypertension (Vascular disorders) | 6 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Constipation (Gastrointestinal disorders) | 4 | 11
Gastritis (Gastrointestinal disorders) | 6 | 8
Eczema (Skin and subcutaneous tissue disorders) | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 15
Periarthritis (Musculoskeletal and connective tissue disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4
Oedema peripheral (General disorders) | 4 | 7
Oedema (General disorders) | 2 | 6
Blood creatine phosphokinase increased (Investigations) | 16 | 15
Brain natriuretic peptide increased (Investigations) | 8 | 6
Blood pressure increased (Investigations) | 0 | 6
Contusion (Injury, poisoning and procedural complications) | 7 | 5
Fall (Injury, poisoning and procedural complications) | 6 | 5

LIMITATIONS AND CAVEATS:
331 participants were randomized in the core phase 2/3 thiazolidine (CCT-004) study and included in the Full Analysis Set in this study. 5 participants from CCT-004 study did not enter this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.